CLINICAL TRIAL: NCT06635265
Title: Single Center Proof-of-Concept Study to Determine the Flow Changes And/or AHI Reduction When Stimulating Two Targets (neural And/or Muscular) for the Treatment of Obstructive Sleep Apnea in Adult Subjects
Brief Title: A Study to Determine the Flow Changes And/or AHI Reduction When Stimulating Two Targets (neural And/or Muscular) for the Treatment of Obstructive Sleep Apnea in Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invicta Medical Inc. (Industry)
Collaborators: Hollywood Private Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM_004
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Disorder
Keywords: Sleep Apnea device
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Electrode arrays placed adjacent to nerves are connected to an external pulse generator to evaluate the effect of short-term stimulation on airflow and/or AHI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Target stimulation (Experimental): Stimulation of a combination of targets: Hypoglossal nerve (HGN) and Ansa Cervicalis (AC), Genioglossus (GG) and AC, HGN and strap muscles, or GG and strap muscles, during an acute and sub-acute phase.
  Interventions: Device: Target Stimulation (HGN, AC, GG, Strap muscles)

INTERVENTIONS:
Device: Target Stimulation (HGN, AC, GG, Strap muscles) — Simulation of a combination of: HGN, AC, GG or strap muscles

SUMMARY:
This Proof-of-Concept study will collect acute and sub-acute flow and/or AHI data following the placement of lead arrays under direct vision. The acute placement and data collection will be collected following the completion of the pre-scheduled neck dissection surgery. The sub-acute data will be collected in a sleep lab during a polysomnography (PSG). Both data collections will be done when stimulating (using an external pulse generator) the hypoglossal nerve or Genioglossus muscle (GG) and a second neural target (Ansa Cervicalis - AC) or the strap muscles (sternohyoid and sternothyroid) with a set of Off-the-Shelf (OTS) electrode arrays.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for inclusion in this study:

* Age above 18 years not under guardianship, under curatorship or under judicial protection.
* Body Mass Index (BMI) < 38 kg/m2.
* Subject must be eligible for neck dissection surgery.
* Written informed consent obtained from the patient prior to performing any study specific procedure.
* Willing and capable to comply with all study requirements, including specific lifestyle considerations, evaluation procedures and questionnaires for the whole duration of the trial.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from participation in this study:

* Major anatomical or functional abnormalities that would impair the ability of the electrode arrays to be positioned.
* Significant comorbidities that contraindicate surgery or general anesthesia.
* Significant tongue weakness.
* Aerodigestive tract tumor or reconstructive surgery performed at the same time as neck dissection.
* Any other chronic medical illness or condition that contraindicates a surgical procedure or general anesthesia in the judgment of the investigator.
* Prior surgery or treatments that could compromise the placement and effectiveness of the electrode array systems:

  * Airway cancer surgery or radiation, or
  * Mandible or maxilla surgery in the previous 3 years (not counting dental treatments).
* Other upper airway surgery to remove obstructions related to OSA in the previous 3 months (e.g., uvulopalatopharyngoplasty (UPPP), tonsillectomy, nasal airway surgery).
* Prior hypoglossal nerve stimulation device implantation.
* Currently pregnant or breastfeeding during the study period.
* Concomitant oral or pharyngeal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Impacts on acute airway opening | Day 0 to 3
  Demonstration of acute airway opening as visually observed under nasoendoscopy when stimulating the HGN or GG and a second target (neural or direct muscle stimulation).
Impacts on airflow during a acute assessment | Day 0 to 3
  Acute increase in airflow when stimulating the HGN or GG and a second target (neural or direct muscle stimulation), measured by changes in amplitude (mA) during target stimulation.

SECONDARY OUTCOMES:
Impacts on airway opening during a sub-acute assessment | Day 0 to 3
  Demonstration of sub-acute flow increase and/or AHI reduction when stimulating two targets simultaneously during natural sleep as measured with polysomnography (PSG), measured by polysomnography.

CONTACTS AND LOCATIONS:
Locations (1):
- Perth Head and Neck Surgery, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No